CLINICAL TRIAL: NCT01739452
Title: National Registry of Patients Diagnosed With Low-risk Myelodysplastic Syndromes According to the Criteria of the WHO / French-American-British Classification System (FAB) and IPSS and Treated With Erythropoietic Agents.
Brief Title: Spanish Registry of Erythropoietic Stimulating Agents Study
Acronym: SPRESAS
Status: Completed | Type: Observational
Sponsor: Grupo Español de Síndromes Mielodisplásicos (Other)
Responsible Party: Sponsor
Other Study IDs: GESMD-SPRESAS-2012-01
Record Dates: First submitted 2012-11-29; First posted 2012-12-03 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2015-04

CONDITIONS: Myelodysplastic Syndrome
Keywords: Low-risk MDS; myelodysplastic syndrome; retrospective
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- erythropoiesis-stimulating agents: Patients diagnosed with low-risk MDS according to IPSS (low or intermediate-1), treated with erythropoiesis-stimulating agents.
- Transfusion support: A control group of patients who received only transfusional support.

SUMMARY:
Reviewing Spanish record of myelodysplastic syndromes (RESMD) data base in the group of patients with MDS. The information will be collected retrospectively from diagnosis of MDS, until the date of December 31, 2011.

DETAILED DESCRIPTION:
Review of RESMD data base in the group of patients with MDS from diagnosis of low risk myelodysplastic syndrome (MDS) and occurrence of anemia that began treatment with erythropoiesis stimulating agent (ESAs) / support transfusional before December 31, 2011. In all cases, data obtained will be prior to the date of the start of the study to ensure its retrospective nature, thus reflecting the routine use of erythropoietic agents in clinical and non-interference in the doctor's clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* The patient has given consent to the collection of data in the RESMD.
* Age ≥ 18 years.
* Patient must be diagnosed with MDS according to WHO classifications or FAB low-risk (IPSS low and intermediate-1) with anemia (Hb ≤ 11 g / dL).
* The patient has studies at the time of diagnosis discard the possibility that MDS anemia is due to deficiency of factors (iron, vitamin B12 or folic acid).
* Initiation of treatment with ESAs or support transfusional at any spanish hematology service before December 31, 2011.

Exclusion Criteria:

* Pretreatment of SMD with hypomethylating agents, lenalidomide, chemotherapy, other.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with MDS according to WHO classifications or FAB low-risk (IPSS low and intermediate-1) with anemia (Hb ≤ 11 g / dL) and treatment (support / ESA) started before December 31, 2011.
Sampling Method: Non-Probability Sample
Enrollment: 722 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Collect and evaluate the Spanish experience of anemia treatment. | 6 months
  Collect and evaluate retrospectively the Spanish experience of anemia treatment in patients diagnosed with low-risk MDS according to IPSS (low or intermediate-1) evaluating the efficacy and safety of treatment with ESAs received for at least 24 weeks and the evolution of a control group of patients who received only transfusional support.

SECONDARY OUTCOMES:
Duration of response | 6 months
  In responders at week 24 of treatment, determine the duration of response after 48 weeks of treatment.
Overall survival. | 6 months
  Evaluate overall survival in the two groups of patients, support transfusional versus ESA.
Adverse events | 6 months
  Security: To determine the frequency, type, intensity and severity of adverse events and their possible relationship with the various ESA and progression to acute myelogenous leukemia.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Consuelo Cañizo, MD, Study Chair — University of Salamanca; María Díez, MD, Study Chair — University of Salamanca